CLINICAL TRIAL: NCT02464904
Title: Pilot Study Evaluating the Effects of Intrapleural Cryotherapy on Tumor Infiltrating Lymphocytes in Malignant Pleural Mesothelioma Using Cryospray Therapy
Brief Title: Intrapleural Cryotherapy for Malignant Pleural Mesothelioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling patients due to enrollment criteria.
Sponsor: Mayo Clinic (Other)
Collaborators: CSA Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Shanda Blackmon, M.D., M.P.H., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-008715
Record Dates: First submitted 2015-05-14; First posted 2015-06-08 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental): Cryospray and biopsies
  Interventions: Procedure: Cryotherapy
- Control (Other): Biopsies
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Cryotherapy — Subjects will have their blood drawn prior to undergoing a staging pleuroscopy. During the pleuroscopy pleural fluid will be collected as well as pleural biopsies (4 to 8 research biopsies). The procedure will involve 2 to 3 applications of cryospray on the location of the disease. After establishing cryofrost over a minimum of a 2 x 2 cm area, cryospray will continue for 15 to 20 seconds, allow a thaw period of 60 seconds followed by one to two repeats in the same location before proceeding onto the next location. We will treat a minimum of 6 x 6 cm area in aggregate. The freezing procedure will be video-recorded and freezing locations and time will be recorded. Approximately, 14 days following the staging pleuroscopy patients will undergo surgical treatment as per standard of care, with repeat blood, pleural fluid and tissue collection.
  Arms: Cryotherapy
Other: Control — Subjects will have their blood drawn prior to undergoing a staging pleuroscopy. During the pleuroscopy pleural fluid will be collected as well as pleural biopsies (4 to 8 research biopsies). Approximately, 14 days following the staging pleuroscopy patients will undergo surgical treatment as per standard of care, with repeat blood, pleural fluid and tissue collection
  Arms: Control

SUMMARY:
Can neoadjuvant intrapleural cryotherapy be safely performed in patients with malignant pleural mesothelioma and will it trigger substantial systemic and local pro-inflammatory changes, resulting in the induction of anti-tumor immunity?

DETAILED DESCRIPTION:
Patients that have been diagnosed, or are suspected of having malignant pleural mesothelioma, a cancer of the pleura, surgery may be considered as an attempt to treat the cancer. As part of the testing needed before surgery, a pleuroscopy or video camera examination of the pleura is necessary to establish the diagnosis and/or to evaluate the extent of the cancer. This study evaluates the effects of cryotherapy (freezing spray) on the ability of a patient's immune system to attack the cancer, as has been reported in other types of cancers. The purpose of this research is to gather information on the safety and effectiveness of cryotherapy in patients with malignant pleural mesothelioma. If successful, this study could provide support for future studies evaluating this new treatment for mesothelioma.

ELIGIBILITY:
Inclusion Criteria

* Subject provides informed consent
* Subject is >18 years of age
* Subject is deemed competent for making medical decisions
* Subject is scheduled to undergo pleuroscopy as part of their standard care for pre-operative clinical staging of malignant pleural mesothelioma
* A negative pregnancy test is required in women of child-bearing potential, as standard of care.
* Subject is mentally capable of understanding study procedures.

Exclusion Criteria

Study subject has any disease or condition that interferes with safe completion of the study including:

* Platelet count < 50K, coagulopathy defined as an International Normalized Ratio (INR) > 1.5
* Anticoagulants such as clopidogrel, heparin, low-molecular weight heparin, warfarin or other novel anticoagulants have not been held for the standard time period published
* Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the surgical or interventional pulmonary attending physicians.
* Hypoxemia with pulse oximetry values <88% or partial pressure of oxygen in arterial blood (PaO2) < 60 on baseline oxygen requirements.
* Concurrent participation in another study involving investigational drugs or investigational medical devices
* Absence of or limited access to the pleural space during medical pleuroscopy.
* Inability to read and understand the necessary study documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07; Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 1 month
  Participants will be monitored for any adverse events that may have resulted from the pleuroscopy procedure.
Mean Number of Tumor Infiltrating Immune Cells as Measured by Immunohistochemistry on Participant Tissue Samples | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Shanda H Blackmon, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials